CLINICAL TRIAL: NCT04407091
Title: A Phase I, Open-Label, Single-Period Study to Assess the Mass Balance Recovery, Pharmacokinetics, Metabolite Profile and Metabolite Identification After Oral Administration of [14C]AZD4831 in Healthy Male Subjects
Brief Title: A Study to Assess the Mass Balance Recovery, Pharmacokinetics, Metabolite Profile and Metabolite Identification of [14C]AZD4831
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6580C00007
Record Dates: First submitted 2020-05-25; First posted 2020-05-29 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Cardiovascular Disease
Keywords: Heart Failure with preserved Ejection Fraction (HFpEF)
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]AZD4831 Oral Solution (Experimental): One 10 mg dose of [14C]AZD4831 Oral Solution
  Interventions: Drug: 14C]AZD4831 Oral Solution

INTERVENTIONS:
Drug: 14C]AZD4831 Oral Solution — 10 mg dose of [14C]AZD4831 Oral Solution
  Other Names: [14C]AZD4831

SUMMARY:
The Sponsor is developing the test medicine, AZD4831, for the potential treatment of cardiovascular disease (CVD). CVD is a general term to describe a range of conditions that affect the heart and blood vessels, examples of CVD include angina (chest pain caused by restricted blood flow to heart muscle) and heart failure (where the heart is unable to pump blood around the body properly). AZD4831 is an inhibitor of a protein that has a role in the formation of fatty deposits in arteries (blood vessels that take blood to the body). It is hoped that by inhibiting this action, AZD4831 will help with the management of CVD.

The study involves radiolabelling (labelling the molecule with radioactive 14C) which is used to locate the molecule within the body. The study will try to assess how much radioactivity can be recovered from the urine and faeces (mass balance recovery) after a single oral dose of [14C]AZD4831. It will also look to identify the breakdown products (metabolites) of the parent drug. It will additionally determine the rate and route of elimination of [14C]AZD4831, along with the level of test medicine in the blood. The safety and tolerability of the test medicine will be assessed. The dose of radiation administered is very low, therefore the risk associated with this is very small.

The study will consist of a single study period involving up to six healthy male volunteers. Up to six male volunteers will receive a dose of 10 mg of the radiolabelled test medicine as an oral solution. Blood, urine and faecal samples will be collected from volunteers whilst they are resident in the clinical unit for up to 336 hours post-dose (Day 15). A follow-up visit will take place seven to ten days after discharge for safety assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated written informed consent prior to any study specific procedures.
2. Healthy male subjects aged 18 to 65 years inclusive at the time of signing informed consent with suitable veins for cannulation or repeated venepuncture.
3. Body mass index (BMI) of 18.0 to 30.0 kg/m2 as measured at screening.
4. Must be willing and able to communicate and participate in the whole study.
5. Must have regular bowel movements (i.e. average stool production of ≥1 and ≤3 stools per day).
6. Must agree to adhere to the contraception requirements

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. History of presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Subjects with uncontrolled or clinically significant thyroid disease as judged by the investigator.
4. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of the IMP.
5. Any clinically significant abnormalities in clinical chemistry, haematology, or urinalysis results, as judged by the investigator. Subjects with known Gilbert's Syndrome or persistently elevated unconjugated bilirubin are not allowed. Subjects with haemoglobin < lower limit of normal (LLN), white blood cell or neutrophil count <LLN (subjects of African origin with neutrophil count <1.8 × 109/L).
6. Any clinically significant abnormal findings in vital signs, as judged by the investigator. Subjects with history of orthostatic hypotension or those who are noted to have a fall in systolic blood pressure >/=20 mmHg or diastolic blood pressure >/=10 mmHg and/or elevation in heart rate of more than 30 bpm or heart rate on standing >120/min when checked 2 min after change of posture at screening or at pre-dose.
7. Any clinically significant abnormalities on 12-lead ECG as judged by the investigator.
8. Any positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C virus antibody, (HCV Ab) and human immunodeficiency virus (HIV) antibody.
9. Known or suspected history of drug abuse within the past 2 years, as judged by the investigator.
10. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the administration of IMP in this study. The period of exclusion ends three months after the final dose or 1 month after the last visit whichever is the longest. Subjects who have done a 14C study in the last 12 months before administration of IMP. Note: subjects consented and screened, but not administered IMP in this study or a previous Phase I study, are not excluded.
11. Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
12. Subjects with ongoing skin disorder or history of significant allergy/hypersensitivity, as judged by the investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD4831 or the formulation excipients. Hay fever is allowed unless it is active.
13. Current smokers or those who have smoked or used nicotine products within the previous 3 months. A confirmed breath carbon monoxide reading of greater than 10 ppm at screening or admission.
14. Current users of e-cigarettes and those who have used e-cigarettes within the last 3 months.
15. Positive screen for drugs of abuse at screening or admission to the clinical unit or positive screen for alcohol at screening or admission to the clinical unit.
16. Known or suspected history of alcohol or drug abuse or excessive intake of alcohol >21 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type)
17. Excessive intake of caffeine-containing drinks or food (e.g. coffee, tea, chocolate) as judged by the investigator. Excessive intake of caffeine defined as the regular consumption of more than 600 mg of caffeine per day (e.g. >5 cups of coffee) or would likely be unable to refrain from the use of caffeine-containing beverages during confinement at the investigational site.
18. Use of drugs or supplements with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
19. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the two weeks prior to administration of investigational product or longer if the medication has a long half life. Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as determined by the investigator.
20. Subjects who are, or are immediate family members of, a study site or sponsor employee.
21. Subjects who have previously received AZD4831.
22. Judgment by the investigator that the subject should not participate in the study if they have any ongoing or recent (i.e. during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements; subjects who have had fever, sore throat or flu like symptoms in the 2 weeks prior to IMP administration.
23. Subjects with pregnant or lactating partners.
24. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study
25. Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance of <80 mL/min using the Cockcroft-Gault equation
26. Vulnerable subjects, e.g. kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order
27. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy male subjects
Enrollment: 8 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-08-06 (Actual)

PRIMARY OUTCOMES:
The cumulative amount of AZD4831 excreted (CumAe) | Urine and faecal samples collected from pre-dose until 336 hours post-dose
  Assessment of the total radioactivity by measuring the cumulative amount of AZD4831 excreted (CumAe)
The cumulative amount of AZD4831 excreted and expressed as a percentage of the administered dose (CumFe) | Urine and faecal samples collected from pre-dose until 336 hours post-dose
  Assessment of the total radioactivity by measuring the cumulative amount of AZD4831 excreted and expressed as a percentage of the administered dose (CumFe)
Assessment of metabolites in plasma by accelerator mass spectrometry (AMS) analysis | Collection of plasma samples from pre-dose until 336 hours post-dose
  Assessment of metabolites and structural identification by AMS analysis
Assessment of metabolites in urine by AMS analysis | Collection of urine samples from pre-dose until 336 hours post-dose
  Assessment of metabolites and structural identification by AMS analysis
Assessment of metabolites in faeces by AMS analysis | Collection of faecal samples from pre-dose until 336 hours post-dose
  Assessment of metabolites and structural identification by AMS analysis

SECONDARY OUTCOMES:
The amount of AZD4831 excreted (Ae) | Collection of urine and faecal samples from pre-dose to 336 hours post-dose.
  Assessment of the rates and routes of elimination by measuring the amount excreted (Ae)
Amount of AZD4831 excreted and expressed as a percentage of the administered dose (Fe) | Collection of urine and faecal samples from pre-dose to 336 hours post-dose
  Assessment of the rates and routes of elimination by measuring the amount excreted and expressing it as a percentage of the administered dose (Fe)
The cumulative amount of AZD4831 excreted (CumAe) | Collection of urine and faecal samples from pre-dose to 336 hours post-dose
  Assessment of the rates and routes of elimination by measuring the cumulative amount excreted (CumAe)
The cumulative amount of AZD4831 excreted and expressed as a percentage of the administered dose (CumFe) | Collection of urine and faecal samples from pre-dose to 336 hours post-dose
  Assessment of the rates and routes of elimination by measuring the cumulative amount excreted and expressed as a percentage of the administered dose (CumFe)
Time to maximum concentration (tmax) for AZD4831 and total radioactivity | Collection of plasma samples from pre-dose to 336 hours post-dose
  Assessment of pharmacokinetics of AZD4831 and total radioactivity by measuring the time to maximum concentration (tmax)
Maximum plasma concentration (cmax) for AZD4831 and total radioactivity | Collection of plasma samples from pre-dose to 336 hours post-dose
  Assessment of pharmacokinetics of AZD4831 and total radioactivity by measuring the maximum concentration (cmax)
Area under the concentration time curve from time zero to the time of the last measureable concentration (AUC0-t) for AZD4831 and total radioactivity | Collection of plasma samples from pre-dose to 336 hours post-dose
  Assessment of pharmacokinetics of AZD4831 and total radioactivity by measuring the concentration time curve from time zero to the last measureable concentration (AUC0-t)
Area under the concentration time curve from time zero to the last quantifiable concentration (AUC0-inf) for AZD4831 and total radioactivity | Collection of plasma samples from pre-dose to 336 hours post-dose
  Assessment of pharmacokinetics of AZD4831 and total radioactivity by measuring the concentration time curve from time zero extrapolated to infinity (AUC0-inf)
Area under the concentration time curve from time of the last measureable concentration to infinity as a percentage of the area under the curve extrapolated to infinity (AUC%extrap) | Collection of plasma samples from pre-dose to 336 hours post-dose
  Assessment of pharmacokinetics of AZD4831 and total radioactivity by measuring the concentration time curve from time of the last measureable concentration to infinity as a percentage of the area under the curve extrapolated to infinity (AUC%extrap)
Apparent terminal elimination half-life (t1/2) for AZD4831 and total radioactivity | Collection of plasma samples from pre-dose to 336 hours post-dose
  Assessment of pharmacokinetics of AZD4831 and total radioactivity by measuring the terminal elimination half-life (t1/2)
First order rate constant associated with the terminal (log-linear) portion of the curve for AZD4831 and total radioactivity | Collection of plasma samples from pre-dose to 336 hours post-dose
  Assessment of pharmacokinetics of AZD4831 and total radioactivity by measuring the first order rate constant associated with the terminal (log-linear) portion of the curve
Total body clearance (CL/F) of AZD4831 and total radioactivity | Collection of plasma samples from pre-dose to 336 hours post-dose
  Assessment of pharmacokinetics of AZD4831 and total radioactivity by measuring total body clearance (CL/F)
Apparent volume of distribution (Vz/F) of AZD4831 and total radioactivity | Collection of plasma samples from pre-dose to 336 hours post-dose
  Assessment of pharmacokinetics of AZD4831 and total radioactivity by measuring the apparent volume of distribution (Vz/F)
Renal clearance (CLR) of AZD4831 in urine | Collection of urine samples from pre-dose to 36 hours post-dose
  Assessment of pharmacokinetics of AZD4831 by measuring renal clearance (CLR)
Evaluation of whole blood to plasma concentration ratios for total radioactivity | Collection of blood samples until 336 hours post-dose
  Assessment of total radioactivity in whole blood and plasma
Number of adverse events (AE) experienced by subjects | AEs recorded from the time of informed consent until discharge from the study (336 hours post-dose)
  Safety and tolerability assessed through the incidence of AEs

OTHER OUTCOMES:
Identification of the chemical structure of major metabolite(s) in plasma | Plasma samples collected until 336 hours post-dose
  Identification of chemical structure of major metabolites of AZD4831
Identification of the chemical structure of major metabolite(s) in urine | Urine samples collected until 336 hours post-dose
  Identification of chemical structure of major metabolites of AZD4831
Identification of the chemical structure of major metabolite(s) in faeces | Faeces samples collected until 336 hours post-dose
  Identification of chemical structure of major metabolites of AZD4831

CONTACTS AND LOCATIONS:
Overall Officials: Somasekhara Menakuru, MBBS, MS, MRCS, DPM, Principal Investigator — Quotient Sciences
Locations (1):
- Research Site, Ruddington, United Kingdom